CLINICAL TRIAL: NCT05731115
Title: A Randomized, Double-blind Clinical Trial to Evaluate the Lot Consistency, Immunogenicity and Safety of 23-valent Pneumococcal Polysaccharide Vaccine in Adults Aged 40-65 Years
Brief Title: Lot-to-lot Consistency of 23-valent Pneumococcal Polysaccharide Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-PPV-4003
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-02

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Vaccine-lot 1 (Experimental): Participants (n=600) aged 40-65 years will receive one dose of 23-valent pneumococcal polysaccharide vaccine of commercial scale production lot 1.
  Interventions: Biological: Experimental 23-valent Pneumococcal
- Experimental Vaccine-lot 2 (Experimental): Participants (n=600) aged 40-65 years will receive one dose of 23-valent pneumococcal polysaccharide vaccine of commercial scale production lot 2.
  Interventions: Biological: Experimental 23-valent Pneumococcal
- Experimental Vaccine-lot 3 (Experimental): Participants (n=600) aged 40-65 years will receive one dose of 23-valent pneumococcal polysaccharide vaccine of commercial scale production lot 3.
  Interventions: Biological: Experimental 23-valent Pneumococcal

INTERVENTIONS:
Biological: Experimental 23-valent Pneumococcal — The investigational vaccine was manufactured by Sinovac Biotech Co., Ltd.25μg each for serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B,17F,18C, 19A, 19F, 20, 22F, 23F, and 33F in 0.5 mL of sodium chloride mixture per injection.

SUMMARY:
This study is a randomized, double-blind phase Ⅳ clinical trial of 23-valent pneumococcal polysaccharide vaccine manufactured by Sinovac Biotech Co., Ltd.The purpose of this study is to evaluate the consistency of three consecutive lots, immunogenicity and safety of 23-valent pneumococcal polysaccharide vaccine of commercial scale in participants aged 40-65 years.

DETAILED DESCRIPTION:
This study is a randomized, double-blind phase Ⅳ clinical trial in subjects aged 40-65 years to evaluate the lot-to-lot consistency,immunogenicity and safety of 23-valent pneumococcal polysaccharide vaccine of commercial scale.The experimental vaccine was manufactured by Sinovac Biotech Co., Ltd.A total of 1800 subjects will be enrolled.The subjects will be randomly divided into three groups in a ratio of 1:1:1 to received one dose of vaccine on day 0.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-65 years in stable health;
* The subjects can understand and voluntarily sign the informed consent form;
* Proven legal identity.

Exclusion Criteria:

* Have received any pneumococcal vaccine;
* History bacterial pneumonia or invasive pneumococcal infectious diseases caused by pneumococci and confirmed by culture;
* Women of childbearing age (menarche to premenopause) are pregnant (including positive urine pregnancy test), breastfeeding or planning pregnancy within 1 month;
* History of asthma, allergy to vaccines or vaccine components, and serious adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema;
* Severe chronic diseases,such as severe cardiovascular diseases, hypertension(Systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg) and diabetes that cannot be controlled by drugs, liver or kidney diseases,malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Autoimmune disease or immune deficiency/immunosuppression;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids(excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* A long history of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs within 30 days prior to receiving the investigational vaccine;
* Receipt of attenuated live vaccines or COVID-19 vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Onset of various acute or chronic diseases within 7 days prior to the study;
* Underarm body temperature before vaccination>37.0°C;
* The subjects participated in other clinical trials during the follow-up period or will be planned to participate other clinical trials within 1 months;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-Geometric Mean Concentration (GMC) | 30 days after vaccination
  GMC for serotype-specific pneumococcal immunoglobulin G (IgG) antibody 30 days after vaccination.

SECONDARY OUTCOMES:
Immunogenicity index-Geometric Mean Increase (GMI) | 30 days after vaccination
  GMI for serotype-specific pneumococcal IgG antibody 30 days after vaccination.
Immunogenicity index-Seroconversion rate (2-fold increase rate) | 30 days after vaccination
  Seroconversion rate (2-fold increase rate) for serotype-specific pneumococcal IgG antibody 30 days after vaccination.
Safety index-Incidence of adverse reactions | Within 30 days after vaccination
  Incidence of adverse reactions within 30 days after vaccination
Safety index-Incidence of adverse reactions | Within 7 days after vaccination
  Incidence of adverse reactions within 7 days after vaccination
Safety index-Incidence of serious adverse events | Within 30 days after vaccination
  Incidence of serious adverse events within 30 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Yunong Zhang, Principal Investigator — Shanxi Provincial Center for Disease Prevention and Control
Locations (2):
- China (2):
  - The First People's Hospital of Yuanping Medical Group, Yuanping, Shanxi
  - Salt Lake District Center for Disease Control and Prevention, Yuncheng, Shanxi

REFERENCES:
- [Derived] Zhang Y, Shi G, Zhou S, Zhao W, Wang L, Li J, Zhao Z, Li G, Geng J, Chen Z, Zhao H, Li Y, Xu L, Wang B, Jiao P, Li G. Lot-to-lot consistency, immunogenicity, and safety of a 23-valent pneumococcal polysaccharide vaccine (PPV23) in healthy adults aged 40-65 years: A randomized, double-blind, controlled, phase IV clinical trial. Hum Vaccin Immunother. 2025 Dec;21(1):2579366. doi: 10.1080/21645515.2025.2579366. Epub 2025 Oct 30. PMID 41165164